CLINICAL TRIAL: NCT03415971
Title: Electromyographic Estimation of Neuro-muscular Coordination of Masticatory Muscles in Patients Treated With Implants (D-2012-057)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North-Western State Medical University named after I.I.Mechnikov (Other)
Responsible Party: Principal Investigator, Silin Alexey Viktorovich, Principal Investigator, North-Western State Medical University named after I.I.Mechnikov
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NWSMU
Record Dates: First submitted 2016-01-28; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Edentulous; Teeth Replacement; Bounded Edentulous Space
MeSH Terms: conditions — Mouth, Edentulous

ARMS (3):
- ASTRA TECH implants (Active Comparator): implant restoration(replace of a missing tooth) - 35 patients
  Interventions: Procedure: EMG befor denture treatment; Procedure: EMG in a month after termination of treatment; Procedure: EMG in a 3 months after termination of treatment
- CROWN (Active Comparator): to fixed denture restorations in own teeth - 32 patients
  Interventions: Procedure: EMG befor denture treatment; Procedure: EMG in a month after termination of treatment; Procedure: EMG in a 3 months after termination of treatment
- non-edontulos (Placebo Comparator): control group will consist 38 non-edotulos patients
  Interventions: Procedure: EMG befor denture treatment

INTERVENTIONS:
Procedure: EMG befor denture treatment
  Other Names: electromyographia
Procedure: EMG in a month after termination of treatment
  Other Names: electromyographia
  Arms: ASTRA TECH implants; CROWN
Procedure: EMG in a 3 months after termination of treatment
  Other Names: electromyographia
  Arms: ASTRA TECH implants; CROWN

SUMMARY:
The result of the study will demonstrate that the functional activity of maxillofacial area with edentulous posterior bounded spaces recovers more effectively in patients treated with restorations on implants comparing to patients treated with fixed dentures.

DETAILED DESCRIPTION:
All patients will be provided with electromyographic research before denture treatment, in a month and three months after the termination of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous bounded space in dental arch (not more that 3 teeth absent)
* Patients ages 20-45 y.o.

Exclusion Criteria:

* Chronical third-degree cardiac failure
* Connective tissue diseases
* Decompensated diabetes
* Neoplastic processes
* Strokes

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
The signals were averaged over 25 ms, with muscle activity assessed as the root mean square (RMS) of the amplitude (µV). sEMG signals were recorded for further analysis. | up to 3 months.
  The present study demonstrated that Osseo Speed implants are safe and reasonable way of treatment for partial tooth loss in the lateral side. There was observed healthy soft tissue and marginal bone stability around the implants. Received data analysis using surface EMG allow to assume than functional state of maxillofacial region and neuromuscular coordination of the muscles of mastication in patients with bounded edentulous space in the lateral side (molars and/or premolars) with implant-supported prosthesis is considerably better than in patients with fixed bridges. Implant-supported prosthesis provide greater bite force for chewing function in comparison with fixed bridges , but certainly less effective than natural teeth. Implant-supported prosthesis increase patients' quality of life and is more convenient for dentoalveolar apparatus.